CLINICAL TRIAL: NCT02087319
Title: Application and Evaluation of PRP on the Therapy for Hair Loss Disorder
Brief Title: Effect of PRP on the Therapy for Hair Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH102-REC1-111
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Hair Loss/Baldness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- platelet-rich plasma (Experimental): hair loss, baldness
  Interventions: Other: hair loss, baldness (patient's own platelet-rich plasma)

INTERVENTIONS:
Other: hair loss, baldness (patient's own platelet-rich plasma) — hair loss, baldness

SUMMARY:
The purpose of study is to examine the advantage of PRP on hair loss and male pattern baldness. The investigators will inject PRP into the scalp regions where with little or no hair, and evaluate the effect and efficiency of PRP on human hair growth.

DETAILED DESCRIPTION:
Hair loss is a disorder in which the hair undergoes aberration growth cycles and falls out from scalp. A number of factors like hormones, genetic factors, diet, endocrine abnormalities, systemic illnesses, drug intake, and hair shaft abnormalities may cause hair loss. Androgen alopecia or male pattern baldness is the most common cause of hair loss caused by progressive shortening of the anagen and increased number of hair follicles in telogen, which has a significant influence on psychological distress.

Except medical treatment and baldness surgery, a new interest in treating hair loss and baldness has been stimulated by using platelet plasma growth factors obtained from the patient's own platelet-rich plasma (PRP). PRP is a portion of plasma fraction of autologous blood having a high concentration of thrombocytes, and can be activated by Thrombin to release multiple growth factors, including platelet-derived growth factor (PDGF), vascular endothelial growth factor (VEGF), epidermal growth factor (EGF), insulin-like growth factor (IGF), and transforming growth factor beta (TGF-β). PRP is known for the capacity to stimulate cell proliferation and differentiation. The action of platelet plasma growth factors on the development of hair follicles has already been established. PRP has also been shown to increase the yield of implanted follicular units during male baldness surgery.

Our study will focus on the advantage of PRP for the treatment of hair loss and male pattern baldness. PRP from autologous blood can be mixed with thrombin in appropriate ratio and inject into the regions on scalp which is interested. We will track and evaluate regularly the effect and efficiency of PRP on human hair growth.

ELIGIBILITY:
Inclusion Criteria:

* patient with hair loss/baldness
* age of 20-70 years old

Exclusion Criteria:

* patient with systemic disorder
* phyco
* patient with coagulation abnormality
* patient with inflammation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
examination the effect of PRP on hair loss/baldness | 1 month
  We will track and evaluate regularly the effect and efficiency of PRP on human hair growing density and newly-formed hair length by phtography and measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Jeng Long-Bin, Study Chair — organ transplantation center
Locations (1):
- China Medical University Hospital, Taichung, Taiwan